CLINICAL TRIAL: NCT04550962
Title: PRospEctiVe charactErization of Asthma Patients Treated With DupilumAb in reaL World Setting
Brief Title: Description of Characteristics, Such as Age, Previous and Concurrent Treatments, Associated Diseases, of Patients With Asthma Treated With Dupilumab (DUPIXENT)
Acronym: REVEAL
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS16688
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — max 1000 characters
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with asthma: Eligible participants are initiating treatment with Dupixent for asthma according to the prescribing information in effect in each country
  Interventions: Drug: Dupilumab SAR231893

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:solution Route of administration: subcutaneous
  Dose regimen:
  Other Names: Dupixent

SUMMARY:
Primary Objective:

The primary objective of the study is to characterize patients initiating DUPIXENT for asthma in a real-world setting, with respect to their medical history, including asthma history and asthma treatment history, socio-demographic, biomarkers (including Fractional exhaled nitric oxide [FeNO]), and concomitant treatments for asthma.

Secondary Objectives:

The secondary objectives of the study are:

* To characterize real-world use patterns of DUPIXENT for asthma (eg, most commonly used regimens, reason for initiation of new asthma treatments, concomitant therapies, treatment durations, and reasons for discontinuation and/or switching)
* To assess the effectiveness of DUPIXENT in asthma patients in a real world setting (lung function improvement, exacerbation rate, asthma control)
* To assess comorbid type 2 conditions (atopic/allergic) and patterns of use and effects of treatment in comorbid conditions in asthma patients treated with Dupixent
* To collect data on HealthCare Resource Utilization (HCRU)
* To collect safety data on study participants in the real-world setting.

DETAILED DESCRIPTION:
Each patient will be followed for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 years or older
* Initiating treatment with Dupixent for asthma according to the country-specific prescribing information
* Willing and able to comply with the required clinic visits, study procedures and assessments.
* Provided signed informed consent

Exclusion Criteria:

* Patients who have a contraindication to Dupixent according to the country-specific prescribing information
* Treatment with Dupixent within 6 months before the baseline visit. Note: for patients who have been treated previously with DUPIXENT a washout period of 6 months is required before Visit 1.
* Any condition that, in the opinion of the Investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from adequately completing the schedule of visits and assessments
* Patients currently participating in any interventional clinical trial which modifies patient care.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with asthma initiating DUPIXENT for their asthma according to the prescribing information in effect in each country.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Characteristics: Socio-demographics | At baseline
  Socio-demographics including but not limited to gender, age, race, weight, and height
Baseline Characteristics: Medical history | At baseline
  Including asthma history and asthma treatment history
Baseline Characteristics: Disease characteristics | At baseline
  Disease characteristics including asthma, comorbid conditions, family history and history of inflammatory diseases
Baseline Characteristics: Biomarkers | At baseline
  Including fractional exhaled nitric oxide (FeNo), blood eosinophils count, immunoglobulin E (IgE total/specific)
Baseline Characteristics: Concomitant treatments for asthma | At baseline

SECONDARY OUTCOMES:
Dupixent and other asthma treatment use patterns | Baseline to Month 36
  Including doses and dose frequency, treatment duration, asthma treatment associations (eg, Dupixent monotherapy, Dupixent + inhaled corticosteroids (ICS), Dupixent + ICS + additional controllers, oral corticosteroid (OCS) burst), and reasons for initiation and for discontinuation/switching.
Lung function | Baseline to Month 36
  Pre and post bronchodilator (BD) forced expiratory volume in 1 second (FEV1) over time.
Annualized exacerbation rate | Baseline to Month 36
  A severe exacerbation event is defined as a deterioration of asthma requiring:
  * Use of systemic corticosteroids for ≥3 days; or
  * Hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.
Patient reported outcomes: Asthma Control Questionnaire (6-item) (ACQ-6) | Baseline to Month 36
  To evaluate asthma control
Patient reported outcomes: Patient Oriented Eczema Measure (POEM) among participants with atopic dermatitis | Baseline to Month 36
  Among participants with atopic dermatitis
Patient reported outcomes: Allergic Rhinitis Visual Analogue Scale (AR-VAS) among participants with allergic rhinitis | Baseline to Month 36
  Among participants with allergic rhinitis
Patient reported outcomes: Sino-nasal Outcome Test (SNOT-22) | Baseline to Month 36
  Among participants with chronic rhinosinusitis with nasal polyps [CRSwNP] and chronic rhinosinusitis [CRS] without nasal polyps [NP])
Healthcare Resource Utilization | Baseline to Month 36
  The Healthcare Resource Utilization (HCRU) collects information on unscheduled healthcare resource encounters including inpatient visits, emergency room visits, physician office visits related to asthma, including the dates of visits and duration of any hospitalizations, together with the reason for the visits
Number of participants with adverse events (AE) and serious adverse events (SAE) | Baseline to Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (41):
- Argentina (6):
  - Investigational Site Number : 0320005, La Plata, Buenos Aires
  - Investigational Site Number : 0320006, Villa Rosa, Buenos Aires
  - Investigational Site Number : 0320001, Ciudad Autonoma Bs As
  - Investigational Site Number : 0320008, Ciudad Autonoma Buenos Aires
  - Investigational Site Number : 0320009, San Miguel de Tucumán
  - Investigational Site Number : 0320004, Santa Fe
- Chile (2):
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Quillota, Región de Valparaíso
- Colombia (3):
  - Investigational Site Number : 1700009, Barranquilla
  - Investigational Site Number : 1700004, Bogotá
  - Investigational Site Number : 1700003, Bucaramanga
- Israel (7):
  - Investigational Site Number : 3760008, Ashdod
  - Investigational Site Number : 3760004, Ashkelon
  - Investigational Site Number : 3760005, Jerusalem
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760001, Kfar Saba
  - Investigational Site Number : 3760006, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
- Investigational Site Number : 4140001, Kuwait City, Kuwait
- Lebanon (3):
  - Investigational Site Number : 4220002, Beirut
  - Investigational Site Number : 4220001, Beirut
  - Investigational Site Number : 4220003, El Achrafiyé
- Investigational Site Number : 4840003, Durango, Mexico
- Investigational Site Number : 6340001, Doha, Qatar
- Russia (6):
  - Investigational Site Number : 6430005, Chelyabinsk
  - Investigational Site Number : 6430007, Moscow
  - Investigational Site Number : 6430004, Moscow
  - Investigational Site Number : 6430006, Rostov-on-Don
  - Investigational Site Number : 6430008, Saratov
  - Investigational Site Number : 6430002, Stavropol
- Saudi Arabia (4):
  - Investigational Site Number : 6820005, Jeddah
  - Investigational Site Number : 6820004, Mecca
  - Investigational Site Number : 6820002, Riyadh
  - Investigational Site Number : 6820001, Riyadh
- Singapore (2):
  - Investigational Site Number : 7020002, Singapore
  - Investigational Site Number : 7020001, Singapore
- United Arab Emirates (5):
  - Investigational Site Number : 7840006, Abu Dhabi
  - Investigational Site Number : 7840007, Dubai
  - Investigational Site Number : 7840001, Dubai
  - Investigational Site Number : 7840004, Sharjah city
  - Investigational Site Number : 7840002, Sharjah city

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org